CLINICAL TRIAL: NCT01594333
Title: A Randomized, Double-blind, Placebo-controlled, Event-driven Trial of Weekly Low-dose Methotrexate (LDM) in the Prevention of Cardiovascular Events Among Stable Coronary Artery Disease Patients With Type 2 Diabetes or Metabolic Syndrome
Brief Title: Cardiovascular Inflammation Reduction Trial
Acronym: CIRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Paul Ridker, Director, Center for Cardiovascular Disease and Prevention, Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012P-000857; U01HL101422 (NIH); U01HL101389 (NIH)
Record Dates: First submitted 2012-05-01; First posted 2012-05-09 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Disease
Keywords: Myocardial Infarction; Stroke; Cardiovascular death; Type 2 Diabetes; Metabolic Syndrome; Cardiovascular Inflammation; Atherothrombosis
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Stroke; Diabetes Mellitus, Type 2; Metabolic Syndrome; Thrombosis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate (Experimental): Methotrexate: Tablet, Oral, Target dose 15-20mg weekly plus 1.0 mg folic acid 6 days/week
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator): Placebo: Tablet, Oral weekly plus 1.0mg folic acid 6 days/week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Tablet, Oral, Target dose 15-20 mg weekly plus 1.0 mg folic acid 6 days/week
  Other Names: Trexall, TEVA Inc (brand of methotrexate)
  Arms: Methotrexate
Drug: Placebo — Tablet, Oral, weekly plus 1.0 mg folic acid 6 days/week
  Arms: Placebo

SUMMARY:
The Cardiovascular Inflammation Reduction Trial (CIRT) is a randomized clinical trial investigating whether taking low-dose methotrexate reduces heart attacks, strokes, or death in people with type 2 diabetes or metabolic syndrome that have had a heart attack or multiple coronary blockages. This trial is funded by the National Heart, Lung, and Blood Institute (NHLBI)/National Institutes of Health (NIH).

DETAILED DESCRIPTION:
While inflammation contributes crucially to atherothrombosis, it is unknown whether inhibition of inflammation per se will lower vascular event rates. The primary aim of the Cardiovascular Inflammation Reduction Trial (CIRT) is to directly test the inflammatory hypothesis of atherothrombosis by evaluating whether or not low-dose methotrexate (LDM) will reduce rates of myocardial infarction, stroke, and cardiovascular death among stable coronary artery disease patients with type 2 diabetes or metabolic syndrome, conditions associated with an enhanced pro-inflammatory response. CIRT is a randomized, double-blind, placebo-controlled, multi-center, event-driven trial that will randomize 7,000 men and women from the United States and Canada. Following a five- to six-week open-label run-in (maximum 8 weeks), eligible participants who have either suffered documented myocardial infarction in the past or have angiographically demonstrated multivessel coronary artery disease in the past will be randomly allocated over a three to four year period to usual care plus placebo or usual care plus LDM. The target methotrexate dose among those allocated to active therapy is 15 to 20 mg po per week, a dose within the range of that commonly used for the treatment of rheumatoid arthritis. All study participants will additionally receive 1.0 mg oral folate to be taken daily six days per week. LDM complications will be minimized through education programs for all investigators and coordinators, through enhanced communication with study participants, by limiting enrollment to those with no evidence of malignancy, hepatitis, renal dysfunction, chronic infection, pulmonary disease, or other risk factors for toxicity; by conducting an initial 5- to 6-week active-therapy run-in (maximum 8 weeks) designed to eliminate individuals who are either intolerant of or unable to adhere to treatment before randomization; and through regular monitoring of liver function and hematologic indices using a centralized methodology designed to ensure participant safety, allow for dose adjustments while maintaining the study blind, and provide an efficient method to address issues of compliance and follow-up on a cost-effective centralized basis. The primary trial endpoint is the rate of myocardial infarction, stroke, or cardiovascular death. Secondary and tertiary endpoints include all-cause mortality, coronary revascularization, incident congestive heart failure, incident peripheral artery disease, incident venous thrombosis, clinically significant aortic stenosis, incident atrial fibrillation, incident diabetes among those with metabolic syndrome but not diabetes at study entry, and hemoglobin A1c (HbA1c) control among those with diabetes at study entry. The trial is event driven such that in the absence of extreme effects, the trial will conclude after accrual of at least 530 primary endpoints, an effect estimated to provide 90 percent power to detect a 25 percent relative risk reduction. The potential clinical impact of CIRT is broad as it has sufficient power to directly address core issues in the inflammatory hypothesis of atherothrombosis, and thus, if successful, will open major new directions for cardiovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at screening
* Documented past history of myocardial infarction OR past evidence of multivessel coronary artery disease by angiography.

  * To qualify on the basis of past history of myocardial infarction, the event must be documented either by hospital records or by evidence on current ECG of Q waves in two contiguous leads and/or an imaging test demonstrating wall motion abnormality or scar. The patient must also have completed any planned coronary revascularization procedures associated with the qualifying event, and be clinically stable for at least 60 days prior to screening.
  * To qualify on the basis of multivessel coronary disease, there must be past angiographic evidence of atherosclerosis in at least 2 major epicardial vessels defined either as the presence of a stent, a coronary bypass graft, or an angiographic lesion of 60% or greater. Left main coronary artery disease that has been revascularized with a stent or bypass graft will qualify as multivessel disease, as will the presence of a 50% or greater isolated left main stenosis. The patient must also have completed any planned coronary revascularization procedures associated with the qualifying event, and be clinically stable for at least 60 days prior to screening.
* History of type 2 diabetes or metabolic syndrome at time of study enrollment
* Willingness to participate as evidenced by signing the study informed consent

Exclusion Criteria:

* Prior history of chronic infectious disease, tuberculosis, or severe fungal disease; chronic hepatitis B or C infection; renal insufficiency; interstitial pneumonitis, bronchiectasis, or pulmonary fibrosis; known chronic pericardial effusion, pleural effusion, or ascites; chronic liver disease; myeloproliferative disorders in the past 5 years; non-basal cell malignancy or treated lymphoproliferative disease within the past 5 years; known HIV positive; life expectancy of < 3 years;
* Chronic inflammatory condition such as lupus or rheumatoid arthritis, ulcerative colitis or Crohn's disease
* White blood cell count < 3,500/ul, hematocrit < 32 percent, or platelet count < 75,000/ul
* Liver transaminase levels (AST or ALT) >upper limit of normal (ULN) or albumin < the lower limit of normal (LLN);
* Creatinine clearance < 40 ml/min as estimated with the Cockcroft-Gault equation;
* History of alcohol abuse or unwillingness to limit alcohol consumption to less than 4 drinks per week
* Women of child bearing potential, even if they are currently using contraception, and women intending to breastfeed.
* Men who plan to father children during the study period or who are unwilling to use effective forms of contraception.
* Requirement for use of drugs that alter folate metabolism (trimethoprim/sulfamethoxazol) or reduce tubular excretion (probenecid) or known allergies to antibiotics making avoidance of trimethoprim impossible;
* Current indication for methotrexate therapy;
* Chronic use of oral steroid therapy or other immunosuppressive or biologic response modifiers. Eligible study participants will be encouraged to have up to date pneumococcal and influenza vaccinations as recommended based on their age and underlying medical conditions.
* Chest X-ray evidence in the past 12 months of interstitial pneumonitis, bronchiectasis, or pulmonary fibrosis. For participants who do not have a chest X-ray in the prior 12 months, a chest X-ray will be obtained at baseline as part of the study protocol.
* New York Heart Association Class IV congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4786 (Actual)
Dates: Start 2013-04; Primary Completion 2019-04-15 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ridker, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (469):
- United States (404):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Appalachian Research Associates, Fort Payne, Alabama
  - Avant Research Associates, LLC, Guntersville, Alabama
  - Saadat Ansari MD LLC, Huntsville, Alabama
  - University of South Alabama: Division of Clinical Research, Mobile, Alabama
  - Heart Vascular of Northern Arizona, Cottonwood, Arizona
  - CardioVascular Associates of Mesa, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, Phoenix, Arizona
  - Scottsdale Medical Imaging, Scottsdale, Arizona
  - The Heart Clinic, Scottsdale, Arizona
  - Pima Heart, Tucson, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Arkansas Cardiology, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Oracle Clinical Research, Inc., Anaheim, California
  - Medical Group of Culver City, Culver City, California
  - Touro University California- Solano County Affiliated Clinics, Fairfield, California
  - University Of California San Francisco, Fresno, California
  - VACCHCS, Fresno, California
  - UCSD Sulpizio Cardiovascular Center, La Jolla, California
  - University Of California San Diego, La Jolla, California
  - Desert Medical Care & Wellness, La Quinta, California
  - Kumar Medical Corporation, Lancaster, California
  - Loma Linda University Health, Loma Linda, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Cardiovascular Innovation and Research, Long Beach, California
  - Los Alamitos Cardiovascular, Los Alamitos, California
  - Faye Montegrande Md. Clinical Research, Los Angeles, California
  - Eastside Clinical Research Associates, Los Angeles, California
  - Salman Khan A. Medical Corporation, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - West LA VA Medical Center, Los Angeles, California
  - VA Northern California Health Care, Mather, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Orange County Heart Institute & Research, Orange, California
  - University of CA Irvine Medical Center, Orange, California
  - Diverse Research Solutions, Oxnard, California
  - Huntington Memorial Hospital, Pasadena, California
  - Central Coast Cardiology, Salinas, California
  - Richard G. Friedman, MD, San Diego, California
  - Ritchken and First MDs, San Diego, California
  - Foundation for Cardiovascular Medicine, San Diego, California
  - San Diego Cardiac Center, San Diego, California
  - Veterans Affairs San Diego Healthcare System, San Diego, California
  - UCSF at Zuckerberg SF General Hospital, San Francisco, California
  - Coastal Heart Medical Group, Inc., Santa Ana, California
  - Comprehensive Cardiovascular Care, Santa Maria, California
  - Pacific Heart and Vascular Medical Group, Stockton, California
  - Manoj D. Aswani M.D., Thousand Oaks, California
  - Touro University California- Solano Public Health Affiliated Clinics, Vallejo, California
  - Munni R. Selagamsetty, Md, Pc, Colorado Springs, Colorado
  - Vijay - Aurora Denver Cardiology, Denver, Colorado
  - Colorado Health Medical Group Heart Center of the Rockies, Fort Collins, Colorado
  - Medical Center of the Rockies Research, Fort Collins, Colorado
  - Unrein - Rocky Vista University Health Center, Parker, Colorado
  - Connecticut Heart and Vascular Center, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Cardiology Physicians/Red Clay Research, Newark, Delaware
  - Boisey Barnes MD, PC, Washington D.C., District of Columbia
  - GWU Medical Faculty Associatin, Inc., Washington D.C., District of Columbia
  - Pianko - Aventura Research Center, LLC, Aventura, Florida
  - North Ridge Heart Associates, Boca Raton, Florida
  - St. Francis Medical Institute, Clearwater, Florida
  - Gonzalez MD & Aswad MD Health Ser, Coral Gables, Florida
  - American Research Institute, Inc., Cutler Bay, Florida
  - Daytona Heart Group, Daytona Beach, Florida
  - Daytona Heart Group, DeLand, Florida
  - Seidman Clinical Trials, Delray Beach, Florida
  - Steven Cohen MD, Delray Beach, Florida
  - Infinite Clinical Research, Doral, Florida
  - International Research Partners, LLC, Doral, Florida
  - Medical Research Institute at Doral, Inc., Doral, Florida
  - Lake Internal Medicine Assocaties, Eustis, Florida
  - Invesclinic, Fort Lauderdale, Florida
  - Primary Care Associates, Fort Myers, Florida
  - Lee Physician Group, Fort Myers, Florida
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Qway Research, Hialeah, Florida
  - State of the Art Research, Hialeah, Florida
  - Healing Touch C&C Research, Hialeah, Florida
  - Luzmed Clinical Research Institute, Hialeah, Florida
  - Viviana Perez MD Research & Cosmetics, Hialeah, Florida
  - Elite Cardiac Research Center LLC, Hialeah, Florida
  - Nova Clinical Research Clinic, Hialeah, Florida
  - Best Quality Research, Inc., Hialeah, Florida
  - South Florida Research Solutions, LLC, Hollywood, Florida
  - John Gutleber Medical Research Office, Homestead, Florida
  - Cardiovascular Medical Associates of Palm Beach, Jupiter, Florida
  - Hope Clinical Research, Kissimmee, Florida
  - SIH Research, LLC, Kissimmee, Florida
  - Medical Research Center of Florida, Miami, Florida
  - LG Diagnostics, Inc., Miami, Florida
  - St. Paul Medical Research Center, Inc., Miami, Florida
  - Team Medical Research, Miami, Florida
  - Paradise Clinical Research, LLC, Miami, Florida
  - GAD Research Center, Miami, Florida
  - Innovation Research Institute, Inc., Miami, Florida
  - Sanitas Research, Miami, Florida
  - Segui - Med Care Research, Miami, Florida
  - South Florida Research Group, LLC, Miami, Florida
  - Vista Health Research, LLC, Miami, Florida
  - D De La Vega MD Research Group, Miami, Florida
  - Lakes Research, LLC, Miami Lakes, Florida
  - Veritas Research Corp., Miami Lakes, Florida
  - Ocean Blue Medical Research Center, Miami Springs, Florida
  - Southwest Florida Research, LLC, Naples, Florida
  - Orlando Healthy Heart Institute, Orlando, Florida
  - Palm Beach Gardens Research Center, LLC, Palm Beach Gardens, Florida
  - Broward Research Center, Pembroke Pines, Florida
  - Pioneer Clinical Research, Pembroke Pines, Florida
  - Sandoval - Broward Research Center, Pembroke Pines, Florida
  - Bay Area Heart Center: 49th Street, St. Petersburg, Florida
  - Bay Area Heart Center: 7th Avenue, St. Petersburg, Florida
  - Lenus Research & Medical Group, Sweetwater, Florida
  - DBC Research, Tamarac, Florida
  - Asclepes Research Centers, Weeki Wachee, Florida
  - Gupta - Premier Heart and Vascular Center, Wesley Chapel, Florida
  - Athens Regional Medical Center, Athens, Georgia
  - Atlanta Veterans Affairs Medical Center, Atlanta, Georgia
  - Laureate Medical Group at Northside, Atlanta, Georgia
  - Synergy Therapeutic Partners, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Atlanta Heart Specialists, LLC, Cumming, Georgia
  - Heart and Rhythm Specialists, Dalton, Georgia
  - Albert F. Johary MD, PC, Dunwoody, Georgia
  - Infinite Clinical Trials, Riverdale, Georgia
  - Atlanta Vanguard Medical Associates, Smyrna, Georgia
  - Herman Clinical Research, LLC, Suwanee, Georgia
  - Atlanta Heart Specialists, LLC, Tucker, Georgia
  - Cardiology Associates of Vidalia, P.C., Vidalia, Georgia
  - VA Pacific Islands Health Care System, Honolulu, Hawaii
  - St. Luke's Idaho Cardiology Associates, Boise, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - Northwest Heart Clinical Research, Arlington Heights, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Med Group-Heart & Vascular Of Illinois, Chicago, Illinois
  - Illinois Heart & Lung Research Center, SC, Normal, Illinois
  - Captain James A. Lovell Federal Health, North Chicago, Illinois
  - Specialty Physicians of Illinois, LLC, Olympia Fields, Illinois
  - Advanced CardioVascular Consultants, Rock Island, Illinois
  - Cardiospecialists, LTD, Dyer, Indiana
  - Martin - Martin Family Practice and Research, Evansville, Indiana
  - Krannert Institute Of Cardiology, Indianapolis, Indiana
  - Community Hospital South, Indianapolis, Indiana
  - Indiana Heart Physicians, Indianapolis, Indiana
  - Medical Consultants, PC, Muncie, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Stahl - Midwest Heart & Vascular Specialists, Overland Park, Kansas
  - Professional Research Network of KS, Wichita, Kansas
  - Robert J. Dole VAMC, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Robley Rex VAMC, Louisville, Kentucky
  - Stoddard - University of Louisville, Louisville, Kentucky
  - Bays - L-MARC Research Center, Louisville, Kentucky
  - Research Integrity LLC, Owensboro, Kentucky
  - Dorothy H. Banish, MD, APMC Study Group, Covington, Louisiana
  - Avant Research Associates, LLC, Crowley, Louisiana
  - North Oaks Cardiology, Hammond, Louisiana
  - American Clinical Research, LLC, Marrero, Louisiana
  - Otis Barnum D.O.P.C., Natchitoches, Louisiana
  - Tulane University Office of Health Research, New Orleans, Louisiana
  - Veterans Affairs Medical Center Shreveport, Shreveport, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Paul A. Shapero, M.D., Bangor, Maine
  - Southern Maine Health Care, Biddeford, Maine
  - InterMed, PA, Portland, Maine
  - Maine Medical Partners Maine Health Cardiology, South Portland, Maine
  - Maine Centers for Healthcare, Westbrook, Maine
  - Sinai Center for Thrombosis Research, Baltimore, Maryland
  - St. Mary's Medical Center, Charlotte Hall, Maryland
  - Calvert Memorial Hospital, Clinton, Maryland
  - Shah Associates, MD, LLC, Prince Frederick, Maryland
  - Peninsula Cardiology Associates, Salisbury, Maryland
  - IRC Clinics, Towson, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - MGH Cardiology, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Massachusetts General Hospital - Chelsea Health Care Center, Chelsea, Massachusetts
  - Pentucket Medical Associates, Inc., Haverhill, Massachusetts
  - VA Central Western Massachusetts Healthca, Leeds, Massachusetts
  - South Shore Internal Medicine, Milton, Massachusetts
  - Lahey Medical Center, Peabody, Massachusetts
  - North Shore Cardiovascular Associates, Salem, Massachusetts
  - Reliant Medical Group, Worcester, Massachusetts
  - Endeavor Medical Research, Alpena, Michigan
  - John D. Dingell Veterans Affairs Medical Center, Detroit, Michigan
  - Trace Research Group at Wayne State University, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Flint Clinical Research, Flint, Michigan
  - Apex Medical Research MI, Inc., Flint, Michigan
  - Garden City Hospital, Garden City, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - National Clinical LLC, Hamtramck, Michigan
  - Academic Cardiology Associates PC, Rochester Hills, Michigan
  - Beaumont Health Center, Royal Oak, Michigan
  - Covenant Medical Center, Inc., Saginaw, Michigan
  - Mid-Michigan Heart & Vascular Center, Saginaw, Michigan
  - Centra Care Heart & Vascular Center at St. Cloud Hospital, Saint Cloud, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Gulfside Clinical Research, LLC, Gulfport, Mississippi
  - University of MS Medical Center, Jackson, Mississippi
  - David M. Headley M.D. PA Planters Clinic, Port Gibson, Mississippi
  - Stern Cardiovascular Foundation, Inc., Southaven, Mississippi
  - Center for Advanced Medicine and Research LLC, Bridgeton, Missouri
  - Center for Advanced Medicine and Research, City of Saint Peters, Missouri
  - Clinical Research Center University of Missouri, Columbia, Missouri
  - Quantum Research LLC, Festus, Missouri
  - Midwest Cardiology Associates, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - VA Medical Center Kansas City, Kansas City, Missouri
  - Lake Regional Cardiovascular Institute, Osage Beach, Missouri
  - CoxHealth: Wheeler Heart & Vascular Center, Springfield, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - VA St. Louis Health Care System (VASTLHCS), St Louis, Missouri
  - SLUCare Cardiology, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Clinical Investigators LLC, St Louis, Missouri
  - Consult and Research Associates, St Louis, Missouri
  - Great Falls Clinic Clinical Research Deptartment, Great Falls, Montana
  - Cone - Montana Medical Research, Missoula, Montana
  - Barrett Clinic, P.C., La Vista, Nebraska
  - Heart Consultants, Omaha, Nebraska
  - Alegent Creighton Health, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Internal Medicine Clinic, Las Vegas, Nevada
  - Red Rock Clinical Research, LLC, Las Vegas, Nevada
  - Sierra Nevada Health Care System, Reno, Nevada
  - Renown Inst for Heart & Vasc Health, Reno, Nevada
  - Lahey Cardiology, Nashua, New Hampshire
  - Family Health at Mount Olive, Flanders, New Jersey
  - Cardiocare, Hillsborough, New Jersey
  - New Jersey Heart, Linden, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Cardiovascular Institute, New Brunswick, New Jersey
  - Palisade Medical Center, North Bergen, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Mercer Bucks Cardiology, Robbinsville, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - Holy Name Medical Center, Inc., Teaneck, New Jersey
  - Total Cardiology Care, LLC, Wayne, New Jersey
  - Westwood Cardiology Associates, Westwood, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Albany Stratton VA Medical Center, Albany, New York
  - Brown - SUNY Downstate Medical Center, Brooklyn, New York
  - Buffalo Heart Group, Buffalo, New York
  - Bassett Healthcare Network, Cooperstown, New York
  - NYU Hudson Valley Cardiology, Cortlandt Manor, New York
  - NYHQ, Flushing, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Long Island Heart Associates, Mineola, New York
  - Winthrop University Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Queens Long Island Medical Group, New Hyde Park, New York
  - Chinatown Cardiology, PC, New York, New York
  - Weill Cornell Medical College and NY Presbyterian, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - DiGiovanna Institute for Medical Education and Research, North Massapequa, New York
  - Champlain Valley Physician Hospital, Plattsburgh, New York
  - Cardiology Associates of Schenectady, Schenectady, New York
  - Novel Research of New York, LLC, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Clinical Study Center of Asheville, Asheville, North Carolina
  - Metrolina Internal Medicine, Charlotte, North Carolina
  - Gaffney Health Services, Charlotte, North Carolina
  - Carolinas Research Center, Charlotte, North Carolina
  - Eastern Carolina Cardiovascular, PA, Elizabeth City, North Carolina
  - Eastern Cardiology, Greenville, North Carolina
  - Northside Clinical Research, Lenoir, North Carolina
  - Lake Shore Clinical Research, LLC., Mooresville, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Cardiology Associates of Carolinas, PA, Morganton, North Carolina
  - Eastern Nephrology Associates, PLLC, New Bern, North Carolina
  - Boice Willis Clinic, Rocky Mount, North Carolina
  - Sanford Cardiology, Sanford, North Carolina
  - Natalie A. Doyle, MD, PA, Wilson, North Carolina
  - Altru Health System Rehab Center, Grand Forks, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Ohio University Heritage College of Osteopathic Medicine, Athens, Ohio
  - Diabetes and Endocrinology Associates of Stark Cit, Canton, Ohio
  - The Lindner Research Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Dayton Heart Center, Dayton, Ohio
  - Dayton Veteran Affairs Medical Center, Dayton, Ohio
  - Colonnade Medical Group, Lancaster, Ohio
  - Middletown Cardiovascular Associates, Middletown, Ohio
  - Comprehensive Heart Care, Inc., Toledo, Ohio
  - Mount Carmel Clinical Cardiovascular Care, Westerville, Ohio
  - Premier Physicians, Westlake, Ohio
  - Wooster Heart Group, Wooster, Ohio
  - Unity Clinical Research, Lindsay, Oklahoma
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Thadani - VA Medical Center Oklahoma City, OK, Oklahoma City, Oklahoma
  - Today Clinical Research, Oklahoma City, Oklahoma
  - Cardiovascular Health Clinic, Oklahoma City, Oklahoma
  - Oklahoma State University Center for Health Sciences, Tulsa, Oklahoma
  - Samaritan Health Services, Corvallis, Oregon
  - Southern Oregon Cardiology, LLC, Medford, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Center for Clinical Res. Abington Health, Abington, Pennsylvania
  - St. Luke's University Hospital, Bethlehem, Pennsylvania
  - Renu-Ca Research Institute, Lower Bucks Hospital, Bristol, Pennsylvania
  - Main Line Health Center, Broomall, Broomall, Pennsylvania
  - Spirit Physician Services, Inc, Camp Hill, Pennsylvania
  - The Chambersburg Hospital, Chambersburg, Pennsylvania
  - Central Bucks Cardiology, Doylestown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Heart Specialists of Lancaster County, Ephrata, Pennsylvania
  - Saint Vincent Consultants in Cardiovascular Diseases, LLC, Erie, Pennsylvania
  - Feasterville Family Healthcare Center, Feasterville, Pennsylvania
  - Christiana Care Health System, Glen Mills, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Harrisburg, Pennsylvania
  - George Isajiw, MD, Lansdowne, Pennsylvania
  - Bucks County Clinical Research, Morrisville, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Lehigh Valley Health Services, Sellersville, Pennsylvania
  - Pish Medical Associates, Inc., Uniontown, Pennsylvania
  - Lehigh Valley Family Practice, Whitehall, Pennsylvania
  - Wilkes-Barre VA Medical Center, Wilkes-Barre, Pennsylvania
  - Partners in Clinical Research, Cumberland, Rhode Island
  - Ocean State Clinical Research Prtnr, Lincoln, Rhode Island
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Ocean State Research Institute, Inc, Providence, Rhode Island
  - South Carolina Heart Center, Columbia, South Carolina
  - Amistad Research Center, LLC, Columbia, South Carolina
  - Miller - SC Internal Medicine Associates.: Irmo, Irmo, South Carolina
  - Charlotte Hearts, Old Point Station, South Carolina
  - Inlet Cardiopulmonary & Associates, Pawleys Island, South Carolina
  - Fusion Clinical Research of Spartanburg, Spartanburg, South Carolina
  - Palmetto Research Center, LLC, Spartanburg, South Carolina
  - New Phase Research & Development, Chattanooga, Tennessee
  - Parkway Medical Group, Fayetteville, Tennessee
  - Stern Cardiovascular Foundation, Inc., Germantown, Tennessee
  - Kore Cardiovascular Research Institutue, Jackson, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - Cardiovascular Research of Knoxville, Knoxville, Tennessee
  - Ramanathan - VAMC Memphis, Memphis, Tennessee
  - Clinical Research Center Meharry Medical College, Nashville, Tennessee
  - Avant Research Associates LLC, Austin, Texas
  - Texas Heart and Vascular Research, LLC, Austin, Texas
  - Southeast TX Clinical Research Center, Beaumont, Texas
  - Cornerstone Family Medicine, Big Spring, Texas
  - IMD Medical Center, Carrollton, Texas
  - Texas Health Physicians Group, Carrollton, Texas
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - North Texas Health Center, Dallas, Texas
  - The Heart Center of Dallas, Dallas, Texas
  - Global Medical Research, DeSoto, Texas
  - The Medical Group of Texas, Fort Worth, Texas
  - Texas Health Physicians Group, Fort Worth, Texas
  - T&R Clinic, P.A., Haltom City, Texas
  - Michele P. Sartori, MD, Houston, Texas
  - Grand Medical Care, Katy, Texas
  - Team Research Of Central Texas, Killeen, Texas
  - Houston Heart and Vascular Associates, Kingwood, Texas
  - Grace Research, LLC, Marshall, Texas
  - Valley Heart Consultants, McAllen, Texas
  - Heart Center, Palo Pinto General Hospital, Mineral Wells, Texas
  - Valley Central Research Inc, Mission, Texas
  - North Hills Medical Research, Inc, North Richland Hills, Texas
  - Grace Research, LLC, Palestine, Texas
  - Avant Research Associates, LLC, Port Arthur, Texas
  - Santoscoy - Health Texas Research Institute, San Antonio, Texas
  - Element Research Group, San Antonio, Texas
  - Schnitzler Cardiovascular Consultants, San Antonio, Texas
  - San Antonio Endovascular & Heart Institute, San Antonio, Texas
  - Acacia Medical Research Institute, Sugar Land, Texas
  - Health Plus Clinical Research, Sugar Land, Texas
  - Lone Star Heart and Vascular Center, Tomball, Texas
  - Northwest Houston Clinical Research, Tomball, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Utah Cardiology, P.C., Layton, Utah
  - Utah Diabetes Center, Salt Lake City, Utah
  - VA Medical Center, White River Junction, White River Junction, Vermont
  - Burke Internal Medicine & Research, Burke, Virginia
  - Seven Corners Medical Research Center, Falls Church, Virginia
  - Hampton Family Practice Research, Hampton, Virginia
  - Tidewater Physicians Multispecialty Group, Hampton, Virginia
  - Virginia Cardiovascular Associates, Manassas, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Tucker Cardiology Associates, P.C., Mechanicsville, Virginia
  - TPMG Clinical Research, Newport News, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Roanoke Heart Institute PLC, Roanoke, Virginia
  - Cardinal Internal Medicine Associates, Woodbridge, Virginia
  - Tidewater Physicians Multispecialty Group, Yorktown, Virginia
  - Frandsen Family Medicine DBA Sound Medi, Port Orchard, Washington
  - Premier Clinical Research, Spokane, Washington
  - Kootenai Heart Clinics, LLC, Spokane, Washington
  - Northside Internal Medicine, Spokane, Washington
  - Northwest Medical Associates, P.S., Vancouver, Washington
  - Cardiology Associates of Bellin Health, Green Bay, Wisconsin
  - Dean Foundation, Madison, Wisconsin
  - University Of Wisconsin, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Columbia St. Mary's, Milwaukee, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (59):
  - The Medical Arts Health Research Group, North Vancouver, British Columbia
  - The Medical Arts Health Research Group, Penticton, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Bramalea Medical Centre, Brampton, Ontario
  - Brampton Research Associates, Brampton, Ontario
  - Philippe R Beaudry Medicine Professional Corporation, Burlington, Ontario
  - Vizel Cardiac Research, Cambridge, Ontario
  - Dr. Linda Sinnaeve's Office, Chatham, Ontario
  - Scisco Clinical Research, Cornwall, Ontario
  - G.S. Cardiac Lab Medicine Professional Corp, Greater Sudbury, Ontario
  - Dr. R. Labonte Professional Med Corp, Greater Sudbury, Ontario
  - Dr. G. Garrioch, Independent Practice, Greater Sudbury, Ontario
  - Dr. Peter Spadafora Health Center, Guelph, Ontario
  - John Stimac, MD, Hamilton, Ontario
  - KMH Cardiology & Diagnostics: Hamilton, Hamilton, Ontario
  - Dr. William Liang, Hamilton, Ontario
  - Source Unique Clinic, Hawkesbury, Ontario
  - Dr. Ronald Fowlis, Kitchener, Ontario
  - University Hospital, London, Ontario
  - Malton Medical Research, Mississauga, Ontario
  - KMH Cardiology & Diagnostics: Mississauga, Mississauga, Ontario
  - Sewa Ram Singal Medicine Professional Corporation, Mississauga, Ontario
  - Newmarket Cardiology Research Group, Newmarket, Ontario
  - Portage Medical Centre, Niagara Falls, Ontario
  - Humber River Regional Hospital, North York, Ontario
  - Bakbak Medicine Professional Corporation, Oshawa, Ontario
  - Dr. James Y. Cha, Oshawa, Ontario
  - University Of Ottawa Heart Institute, Ottawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Steeple Hill Medical Centre, Pickering, Ontario
  - Sarnia Institute Of Clinical Research, Sarnia, Ontario
  - Scarborough Cardiology Research, Scarborough Village, Ontario
  - Scarborough General Hospital Cardiology Research Associates, Scarborough Village, Ontario
  - Milliken Medical Centre, Scarborough Village, Ontario
  - Canadian Centre for Research on Diabetes, Smith Falls, Ontario
  - Lake Shore Cardiology, St. Catharines, Ontario
  - Sardar Medical Clinic, St. Thomas, Ontario
  - Dr. Laurence Gibbs Medicine Professional Corp., Thedford, Ontario
  - Tillsonburg Medical Centre, Tillsonburg, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Weston Road Medical Clinic, Toronto, Ontario
  - Dr. Nigel Jagan Medicine Professional Corporation, Whitby, Ontario
  - Dr. Nwadiaro Medicine Professional Corp, Windsor, Ontario
  - Viacar Recherche Clinique Inc., Brossard, Quebec
  - Ecogene-21, Chicoutimi, Quebec
  - Q&T Research Chicoutimi, Chicoutimi, Quebec
  - Viacar Recherche Clinique Inc., Greenfield Park, Quebec
  - CHUM Hotel-Dieu, Montreal, Quebec
  - Recherche Clinique Sigma, Inc., Québec, Quebec
  - Iucpq, Québec, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec
  - CardioVasc HR, Saint-Jean-sur-Richelieu, Quebec
  - ViaCar Recherche Clinique Inc, Saint-Lambert, Quebec
  - Viacar Recherche Clinique, Saint-Lambert, Quebec
  - Hopital Pierre-Le Gardeur, Terrebonne, Quebec
- Puerto Rico (6):
  - Instituto Sanacoop, Bayamón
  - San Juan Bautista School of Medicine, Caguas
  - Norma S. Severino-Pacheco, MD, Canovanas
  - Cardiometabolic Research Center, Ponce
  - Miguel Sosa-Padilla, MD, San Juan
  - Yolanda Sierra Quinones, MD, Toa Baja

REFERENCES:
- [Derived] Cui J, Ridker PM, Solomon DH. Blood pressure changes during methotrexate treatment: results from a randomized placebo-controlled trial among patients with cardiovascular risk. Rheumatology (Oxford). 2025 Jun 1;64(6):3917-3920. doi: 10.1093/rheumatology/keae604. PMID 39657237
- [Derived] Cui J, Chasman DI, Raychaudhuri S, Xu C, Ridker PM, Solomon DH, Karlson EW. Genetics are not likely to offer clinically useful predictions for elevated liver enzyme levels in patients using low dose methotrexate. Semin Arthritis Rheum. 2022 Aug;55:152036. doi: 10.1016/j.semarthrit.2022.152036. Epub 2022 May 28. PMID 35671649
- [Derived] Reiss AB, Teboul I, Kasselman L, Ahmed S, Carsons SE, De Leon J. Methotrexate effects on adenosine receptor expression in peripheral monocytes of persons with type 2 diabetes and cardiovascular disease. J Investig Med. 2022 Aug;70(6):1433-1437. doi: 10.1136/jim-2022-002355. Epub 2022 May 23. PMID 35606100
- [Derived] Sparks JA, Vanni KMM, Sparks MA, Xu C, Santacroce LM, Glynn RJ, Ridker PM, Solomon DH. Effect of Low-Dose Methotrexate on eGFR and Kidney Adverse Events: A Randomized Clinical Trial. J Am Soc Nephrol. 2021 Dec 1;32(12):3197-3207. doi: 10.1681/ASN.2021050598. Epub 2021 Dec 1. PMID 34551998
- [Derived] Xu C, Selhub J, Jacques P, Paynter NP, MacFadyen JG, Glynn RJ, Ridker PM, Solomon DH. Adverse effects related to methotrexate polyglutamate levels: adjudicated results from the cardiovascular inflammation reduction trial. Rheumatology (Oxford). 2021 Jun 18;60(6):2963-2968. doi: 10.1093/rheumatology/keaa650. PMID 34144603
- [Derived] Sparks JA, Dellaripa PF, Glynn RJ, Paynter NP, Xu C, Ridker PM, Solomon DH. Pulmonary Adverse Events in Patients Receiving Low-Dose Methotrexate in the Randomized, Double-Blind, Placebo-Controlled Cardiovascular Inflammation Reduction Trial. Arthritis Rheumatol. 2020 Dec;72(12):2065-2071. doi: 10.1002/art.41452. Epub 2020 Oct 7. PMID 32741143
- [Derived] Ridker PM, MacFadyen JG, Glynn RJ, Bradwin G, Hasan AA, Rifai N. Comparison of interleukin-6, C-reactive protein, and low-density lipoprotein cholesterol as biomarkers of residual risk in contemporary practice: secondary analyses from the Cardiovascular Inflammation Reduction Trial. Eur Heart J. 2020 Aug 14;41(31):2952-2961. doi: 10.1093/eurheartj/ehaa160. PMID 32221587
- [Derived] Solomon DH, Glynn RJ, Karlson EW, Lu F, Corrigan C, Colls J, Xu C, MacFadyen J, Barbhaiya M, Berliner N, Dellaripa PF, Everett BM, Pradhan AD, Hammond SP, Murray M, Rao DA, Ritter SY, Rutherford A, Sparks JA, Stratton J, Suh DH, Tedeschi SK, Vanni KMM, Paynter NP, Ridker PM. Adverse Effects of Low-Dose Methotrexate: A Randomized Trial. Ann Intern Med. 2020 Mar 17;172(6):369-380. doi: 10.7326/M19-3369. Epub 2020 Feb 18. PMID 32066146
- [Derived] Ridker PM, Everett BM, Pradhan A, MacFadyen JG, Solomon DH, Zaharris E, Mam V, Hasan A, Rosenberg Y, Iturriaga E, Gupta M, Tsigoulis M, Verma S, Clearfield M, Libby P, Goldhaber SZ, Seagle R, Ofori C, Saklayen M, Butman S, Singh N, Le May M, Bertrand O, Johnston J, Paynter NP, Glynn RJ; CIRT Investigators. Low-Dose Methotrexate for the Prevention of Atherosclerotic Events. N Engl J Med. 2019 Feb 21;380(8):752-762. doi: 10.1056/NEJMoa1809798. Epub 2018 Nov 10. PMID 30415610
- [Derived] Everett BM, Pradhan AD, Solomon DH, Paynter N, Macfadyen J, Zaharris E, Gupta M, Clearfield M, Libby P, Hasan AA, Glynn RJ, Ridker PM. Rationale and design of the Cardiovascular Inflammation Reduction Trial: a test of the inflammatory hypothesis of atherothrombosis. Am Heart J. 2013 Aug;166(2):199-207.e15. doi: 10.1016/j.ahj.2013.03.018. Epub 2013 May 3. PMID 23895801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9321 subjects were screened and 4786 subjects were randomized starting from April, 2013 through March 2018 in 417 clinical sites in Canada and the United States
Pre-assignment Details: 9321 subjects were screened, 2987 were found to be ineligible and 176 were discontinued due to premature trial closure prior to entering the open label run-in. 6158 started the run-in. Of those, 1171 were ineligible, 201 were discontinued due to premature trial closure and 4786 subjects were randomly assigned to either Methotrexate or Placebo
Period: Overall Study
Arm/Group | Methotrexate | Placebo
Started | 2391 | 2395
Completed | 2230 | 2244
Not Completed | 161 | 151
Not completed — Death | 96 | 83
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 60 | 63

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Placebo | Total
Number analyzed (Participants) | 2391 | 2395 | 4786
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age at randomization
  years | 65.6 [59.7 to 71.8] | 66.0 [59.8 to 71.7] | 65.8 [59.7 to 71.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 461 | 437 | 898
  Male | 1930 | 1958 | 3888
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 206 | 177 | 383
  White/Non-hispanic or Latino | 1801 | 1837 | 3638
  Asian | 89 | 92 | 181
  Black or African American | 186 | 152 | 338
  American Indian or Alaska Native | 6 | 6 | 12
  Native Hawaiian or other Pacific Islander | 3 | 6 | 9
  Multiracial | 13 | 7 | 20
  Other | 42 | 45 | 87
  White, Unknown Ethnicity | 45 | 73 | 118
Region of Enrollment [Number; unit: participants]
  Canada | 407 | 404 | 811
  Puerto Rico | 19 | 17 | 36
  United States | 1965 | 1974 | 3939
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 267 | 270 | 537
  Past smoker | 1173 | 1215 | 2388
  Never smoked cigarettes | 951 | 910 | 1861
Alcohol use [Count of Participants; unit: Participants]
  Rarely/Never | 1487 | 1473 | 2960
  <=1 drink/week | 514 | 520 | 1034
  >1 drink/week | 390 | 402 | 792
Body Mass Index [Median (Inter-Quartile Range); unit: kilograms per meter squared] | 31.6 [28.2 to 35.5] | 31.3 [28.1 to 35.6] | 31.5 [28.2 to 35.6]
History of diagnosed hypertension [Count of Participants; unit: Participants] — Population: One subject is missing this information
  Participants
    number analyzed (Participants) | 2391 | 2394 | 4785
    Yes | 2153 | 2169 | 4322
    No | 238 | 225 | 463
Qualifying event [Count of Participants; unit: Participants]
  Myocardial infarction | 1451 | 1458 | 2909
  Multivessel coronary disease | 940 | 937 | 1877
Qualifying coexisting condition [Count of Participants; unit: Participants]
  Diabetes only | 788 | 823 | 1611
  Metabolic syndrome only | 771 | 780 | 1551
  Diabests and metabolic syndrome | 832 | 792 | 1624
History of congestive heart failure [Count of Participants; unit: Participants] — Population: One subject is missing this information
  Participants
    number analyzed (Participants) | 2391 | 2394 | 4785
    Yes | 288 | 332 | 620
    No | 2103 | 2062 | 4165
History of percutaneous coronary intervention [Count of Participants; unit: Participants] — Population: One subject is missing this information
  Participants
    number analyzed (Participants) | 2391 | 2394 | 4785
    Yes | 1396 | 1420 | 2816
    No | 995 | 974 | 1969
History of coronary-artery bypass grafting [Count of Participants; unit: Participants] — Population: One subject is missing this information
  Participants
    number analyzed (Participants) | 2391 | 2394 | 4785
    Yes | 1010 | 1032 | 2042
    No | 1381 | 1362 | 2743
Family history of premature myocardial infarction [Count of Participants; unit: Participants] — A family history of premature myocardial infarction was considered to be an event occurring in the mother before the age of 65 or in the father before the age of 55. Population: 552 subjects are missing this information
  Participants
    number analyzed (Participants) | 2118 | 2116 | 4234
    Yes | 550 | 536 | 1086
    No | 1568 | 1580 | 3148
Family history of premature stroke [Count of Participants; unit: Participants] — A family history of premature stroke infarction was considered to be an event occurring in the mother before the age of 65 or in the father before the age of 55. Population: 482 subjects are missing this information
  Participants
    number analyzed (Participants) | 2144 | 2160 | 4304
    Yes | 142 | 136 | 278
    No | 2002 | 2024 | 4026
Use of ACE inhibitor or ARB [Count of Participants; unit: Participants] — ACE denotes angiotensin-converting enzyme and ARB denotes angiotensin-receptor blocker
  Participants
    Yes | 1736 | 1724 | 3460
    No | 655 | 671 | 1326
Use of a statin [Count of Participants; unit: Participants]
  Yes | 2058 | 2052 | 4110
  No | 333 | 343 | 676
Use of a beta-blocker [Count of Participants; unit: Participants]
  Yes | 1870 | 1905 | 3775
  No | 521 | 490 | 1011
Use of antiplatelet or antithrombotic agent [Count of Participants; unit: Participants]
  Yes | 2082 | 2054 | 4136
  No | 309 | 341 | 650
Total cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Values are from enrollment, before the active-treatment run-in phase Population: 45 subjects are missing this information
  mg/dL
    number analyzed (Participants) | 2369 | 2372 | 4741
    (all) | 141.0 [122.0 to 168.0] | 140.9 [122.0 to 164.0] | 141.0 [122.0 to 166.0]
Low density lipoprotein cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Values are from enrollment, before the active-treatment run-in phase Population: 192 subjects are missing this information
  mg/dL
    number analyzed (Participants) | 2288 | 2306 | 4594
    (all) | 68.0 [54.0 to 87.0] | 68.0 [53.3 to 86.0] | 68.0 [53.7 to 87.0]
High density lipoprotein cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Values are from enrollment, before the active-treatment run-in phase Population: 45 subjects are missing this information
  mg/dL
    number analyzed (Participants) | 2369 | 2372 | 4741
    (all) | 41.0 [34.7 to 49.0] | 41.0 [35.0 to 48.0] | 41.0 [35.0 to 48.0]
Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] — Values are from enrollment, before the active-treatment run-in phase Population: 45 subjects are missing this information
  mg/dL
    number analyzed (Participants) | 2369 | 2372 | 4741
    (all) | 135.4 [98.0 to 191.2] | 136.0 [98.2 to 191.6] | 135.4 [98.0 to 191.2]
High-sensitivity C-reactive protein level [Median (Inter-Quartile Range); unit: mg/liter] — Values are from enrollment, before the active-treatment run-in phase Population: 95 subjects are missing this information
  mg/liter
    number analyzed (Participants) | 2343 | 2348 | 4691
    (all) | 1.53 [0.78 to 3.59] | 1.50 [0.70 to 3.29] | 1.51 [0.74 to 3.44]
Glycated hemoglobin level [Median (Inter-Quartile Range); unit: %] — Values are from enrollment, before the active-treatment run-in phase Population: 36 subjects are missing this information
  %
    number analyzed (Participants) | 2372 | 2378 | 4750
    (all) | 6.6 [6.0 to 7.5] | 6.5 [5.9 to 7.5] | 6.5 [6.0 to 7.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Major Adverse Cardiovascular Events
Description: The first occurrence of Major Adverse Cardiovascular Event which is defined as the occurrence of one or more of the following: Cardiovascular Death, Non-Fatal Myocardial Infarction or Non-Fatal Stroke.
Time Frame: From randomization to trial end (April 2, 2018) up to a maximum of 5 years
Population: All randomized subjects
Measure: Number; unit: participants
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 2391 | 2395
participants | 170 | 167
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; Test type: Superiority; p = 0.91, Log Rank — 2-sided unadjusted p-value; Stratified according to type of qualifying event, time of qualifying event and risk status(diabetes or metabolic syndrome alone); Cox Proportional Hazard = 1.01, 95% CI 2-sided [0.82 to 1.25] — Confidence intervals have not been adjusted for multiplicity, and therefore inferences drawn from these intervals may not be reproducible

2. Primary Outcome: Number of Subjects With Major Adverse Cardiovascular Event or Hospitalization for Unstable Angina That Led to Urgent Coronary Revascularization
Description: The first occurrence of Major Adverse Cardiovascular Event or Hospitalization for Unstable Angina that led to Urgent Coronary Revascularization.
Time Frame: From randomization to trial end (April 2, 2018) - up to a maximum of 5 years
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 2391 | 2395
participants | 201 | 207
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; Test type: Superiority; p = 0.67, Log Rank — 2-sided unadjusted p-value; Stratified according to type of qualifying event, time of qualifying event and risk status(metabolic syndrome alone or diabetes at enrollment); Cox Proportional Hazard = 0.96, 95% CI 2-sided [0.79 to 1.16] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Subjects With All-cause Mortality
Description: Subjects who died from any cause.
Time Frame: From randomization to the trial end (April 2, 2018) up to a maximum of 5 years
Population: All Randomized Participants
Measure: Number; unit: participants
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 2391 | 2395
participants | 96 | 83
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; Test type: Superiority; p = 0.32, Log Rank — 2-sided unadjusted p-value; Stratified according to type of qualifying event, time of qualifying event and risk status (metabolic syndrome alone or diabetes at enrollment); Cox Proportional Hazard = 1.16, 95% CI 2-sided [0.87 to 1.56] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Subjects With Major Adverse Cardiovascular Event or Any Coronary Revascularization
Description: The first occurrence of Major Adverse Cardiovascular Event or Any Coronary Revascularization.
Time Frame: From randomization to the trial end (April 2, 2018) - up to a maximum of 5 years
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 2391 | 2395
participants | 278 | 288
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; Test type: Superiority; p = 0.57, Log Rank — 2-sided unadjusted p-value; Stratified according to type of qualifying event, time of qualifying event and risk status (metabolic syndrome alone or diabetes) at enrollment; Cox Proportional Hazard = 0.95, 95% CI 2-sided [0.81 to 1.12] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Subjects With Hospitalization for Congestive Heart Failure
Description: The first occurrence of Hospitalization for Congestive Heart Failure
Time Frame: From randomization to trial end (April 2, 2018) up to a maximum of 5 years
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 2391 | 2395
participants | 48 | 53
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; Test type: Superiority; p = 0.54, Log Rank — 2-sided unadjusted p-value; Stratified according to type of qualifying event, type of qualifying event and risk status (diabetes or metabolic syndrome alone) at enrollment; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.60 to 1.31] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Subjects With Major Adverse Cardiovascular Event, Coronary Revascularization, Hospitalization for Congestive Heart Failure or All Cause Mortality
Description: The first occurrence of Major Adverse Cardiovascular Event, Coronary Revascularization, Hospitalization for Congestive Heart Failure or All Cause Mortality.
Time Frame: From randomization to trial end (April 2, 2018) up to a maximum of 5 years
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 2391 | 2395
participants | 344 | 345
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; Test type: Superiority; p = 0.80, Log Rank — 2-sided unadjusted p-value; Stratified according to type of qualifying event, time since qualifying event and risk status (diabetes or metabolic syndrome alone) at enrollment; Cox Proportional Hazard = 0.98, 95% CI 2-sided [0.84 to 1.14] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Subjects With New Onset Type 2 Diabetes
Description: New onset type 2 diabetes among those without diabetes at baseline. Baseline diabetes is defined as any of the following prior to randomization: clinician report of diabetes, use of antidiabetic medication, hbA1c >=6.5 or fasting plasma glucose >=126.
Time Frame: From randomization to the trial end (April 2, 2018) - up to 5 years
Population: Randomized participants without pre-randomization diabetes
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 605 | 620
Participants | 4 | 6

8. Other Pre Specified Outcome: Number of Subjects With Hospitalization for Unstable Angina That Led to Unplanned Coronary Revascularization
Description: The first occurrence of hospitalization for unstable angina that led to unplanned coronary revascularization
Time Frame: From randomization to the trial end (April 2, 2018) up to 5 years
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 2391 | 2395
participants | 41 | 50
Statistical Analysis 1: Comparison: Methotrexate; Test type: Superiority; p = 0.31, Log Rank — 2-sided unadjusted p-value; Stratified according to type of qualifying event, time of qualifying event and risk status (diabetes or metabolic syndrome alone) at enrollment; Cox Proportional Hazard = 0.81, 95% CI 2-sided [0.53 to 1.22] — [estimate comment as in outcome 1, analysis 1]

9. Other Pre Specified Outcome: Number of Subjects With Coronary Revascularization
Description: The first occurrence of coronary revascularization
Time Frame: From randomization to trial end (April 2, 2018) up to 5 years
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 2391 | 2395
participants | 190 | 205
Statistical Analysis 1: Comparison: Methotrexate vs Placebo; Test type: Superiority; p = 0.38, Log Rank — 2-sided unadjusted p-value; [statistical method as in outcome 8, analysis 1]; Cox Proportional Hazard = 0.92, 95% CI 2-sided [0.75 to 1.12] — [estimate comment as in outcome 1, analysis 1]

10. Other Pre Specified Outcome: Number of Subjects With Peripheral Artery Disease
Description: The first occurrence of new or worsening of peripheral artery disease
Time Frame: From randomization to the trial end (April 2, 2018) - up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number of Subjects With Deep Vein Thrombosis or Pulmonary Embolism
Description: The first occurrence of symptomatic deep vein thrombosis or pulmonary embolism
Time Frame: From randomization to the trial end (April 2, 2018) - up to 5 years
Population: The trial was ended prematurely. There were not sufficient outcome measures for analysis
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Number of Subjects With Aortic Stenosis
Description: The first occurrence of clinically significant aortic stenosis
Time Frame: From randomization to the trial end (April 2, 2018) - up to 5 years
Population: The trial ended prematurely. There were not sufficient outcome measures for analysis.
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Number of Subjects With Atrial Fibrillation
Description: The first occurrence of new or worsening of atrial fibrillation
Time Frame: From randomization to the trial end (April 2, 2018) - up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From randomization to the trial end (April 2, 2018) - up to 5 years.
Description: Pre-specified adverse events were collected via questions on the case report forms (CRFs) at each visit. Sites queried participants about any other adverse events and recorded them using a standard adverse event form that included the seriousness, relatedness, severity and outcomes. Those adverse events were MedDRA coded.
Arm/Group | Methotrexate | Placebo
All-Cause Mortality (participants affected / at risk) | 96/2391 | 83/2395
Serious Adverse Events (participants affected / at risk) | 569/2391 | 549/2395
Other Adverse Events (participants affected / at risk) | 1488/2391 | 1399/2395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=2391) | Placebo (N=2395)
Pneumonia (Infections and infestations) | 29 | 28
Cellulitis (Infections and infestations) | 19 | 15
Urinary tract infection (Infections and infestations) | 12 | 9
Sepsis (Infections and infestations) | 12 | 7
Infection (Infections and infestations) | 6 | 7
Diverticulitis (Infections and infestations) | 4 | 8
Bronchitis (Infections and infestations) | 7 | 2
Osteomyelitis (Infections and infestations) | 8 | 1
Gastroenteritis (Infections and infestations) | 2 | 4
Influenza (Infections and infestations) | 1 | 4
Localised infection (Infections and infestations) | 4 | 0
Pyelonephritis (Infections and infestations) | 1 | 3
Septic shock (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Appendicitis (Infections and infestations) | 0 | 3
Bacteraemia (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 3
Urosepsis (Infections and infestations) | 1 | 2
Abdominal wall abscess (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 2
Bacterial disease carrier (Infections and infestations) | 1 | 1
Bronchitis viral (Infections and infestations) | 1 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 2
Groin abscess (Infections and infestations) | 1 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 2
Perirectal abscess (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 2
Abscess (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis shigella (Infections and infestations) | 1 | 0
Genital herpes (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lyme disease (Infections and infestations) | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 10
Abdominal pain (Gastrointestinal disorders) | 9 | 6
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Pancreatitis acute (Gastrointestinal disorders) | 2 | 3
Intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Retroperitoneal mass (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 24 | 16
Transient ischaemic attack (Nervous system disorders) | 9 | 9
Dizziness (Nervous system disorders) | 6 | 3
Presyncope (Nervous system disorders) | 4 | 2
Convulsion (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 3 | 2
Dysarthria (Nervous system disorders) | 2 | 2
Dementia (Nervous system disorders) | 1 | 2
Encephalopathy (Nervous system disorders) | 1 | 2
Hemiparesis (Nervous system disorders) | 2 | 1
Migraine (Nervous system disorders) | 1 | 2
VIIth nerve paralysis (Nervous system disorders) | 0 | 2
Aphasia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Clonus (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 1
Neuromyopathy (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Paresis (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Radicular pain (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 0 | 1
Chest pain (General disorders) | 76 | 67
Non-cardiac chest pain (General disorders) | 8 | 3
Chest discomfort (General disorders) | 4 | 3
Pyrexia (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 0 | 4
Asthenia (General disorders) | 3 | 0
Systemic inflammatory response syndrome (General disorders) | 2 | 0
Adverse event (General disorders) | 1 | 0
Device malfunction (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Medical device complication (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Organ failure (General disorders) | 0 | 1
Swelling (General disorders) | 0 | 1
Ulcer haemorrhage (General disorders) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 10 | 11
Hospitalisation (Surgical and medical procedures) | 4 | 6
Hip arthroplasty (Surgical and medical procedures) | 6 | 3
Surgery (Surgical and medical procedures) | 2 | 7
Spinal laminectomy (Surgical and medical procedures) | 3 | 4
Gastrectomy (Surgical and medical procedures) | 3 | 3
Implantable defibrillator insertion (Surgical and medical procedures) | 3 | 2
Cardiac pacemaker insertion (Surgical and medical procedures) | 4 | 0
Hip surgery (Surgical and medical procedures) | 2 | 2
Knee operation (Surgical and medical procedures) | 3 | 1
Toe amputation (Surgical and medical procedures) | 2 | 2
Cardiac ablation (Surgical and medical procedures) | 1 | 2
Carotid endarterectomy (Surgical and medical procedures) | 1 | 2
Gallbladder operation (Surgical and medical procedures) | 2 | 1
Joint arthroplasty (Surgical and medical procedures) | 2 | 1
Shoulder arthroplasty (Surgical and medical procedures) | 2 | 1
Aortic valve replacement (Surgical and medical procedures) | 0 | 2
Cardioversion (Surgical and medical procedures) | 2 | 0
Colectomy (Surgical and medical procedures) | 2 | 0
Gastric bypass (Surgical and medical procedures) | 1 | 1
Intervertebral disc operation (Surgical and medical procedures) | 2 | 0
Mitral valve repair (Surgical and medical procedures) | 2 | 0
Nephrectomy (Surgical and medical procedures) | 0 | 2
Penile prosthesis insertion (Surgical and medical procedures) | 2 | 0
Shoulder operation (Surgical and medical procedures) | 2 | 0
Stent placement (Surgical and medical procedures) | 0 | 2
Tooth extraction (Surgical and medical procedures) | 1 | 1
Abdominal hernia repair (Surgical and medical procedures) | 1 | 0
Ankle operation (Surgical and medical procedures) | 0 | 1
Aortic aneurysm repair (Surgical and medical procedures) | 0 | 1
Appendicectomy (Surgical and medical procedures) | 1 | 0
Bladder neoplasm surgery (Surgical and medical procedures) | 0 | 1
Cancer surgery (Surgical and medical procedures) | 1 | 0
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 0 | 1
Cataract operation (Surgical and medical procedures) | 1 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Craniotomy (Surgical and medical procedures) | 0 | 1
Finger amputation (Surgical and medical procedures) | 0 | 1
Fistula repair (Surgical and medical procedures) | 0 | 1
Foot amputation (Surgical and medical procedures) | 1 | 0
Hernia repair (Surgical and medical procedures) | 0 | 1
Implantable defibrillator replacement (Surgical and medical procedures) | 0 | 1
Intestinal resection (Surgical and medical procedures) | 1 | 0
Lung lobectomy (Surgical and medical procedures) | 1 | 0
Mastectomy (Surgical and medical procedures) | 0 | 1
Oesophagectomy (Surgical and medical procedures) | 1 | 0
Oesophagogastric fundoplasty (Surgical and medical procedures) | 1 | 0
Partial lung resection (Surgical and medical procedures) | 0 | 1
Pelvic floor repair (Surgical and medical procedures) | 0 | 1
Prolapse repair (Surgical and medical procedures) | 1 | 0
Prostatectomy (Surgical and medical procedures) | 0 | 1
Radical cystectomy (Surgical and medical procedures) | 0 | 1
Radiotherapy (Surgical and medical procedures) | 1 | 0
Removal of internal fixation (Surgical and medical procedures) | 0 | 1
Retinopexy (Surgical and medical procedures) | 1 | 0
Small intestinal resection (Surgical and medical procedures) | 0 | 1
Spinal cord operation (Surgical and medical procedures) | 0 | 1
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 1 | 0
Umbilical hernia repair (Surgical and medical procedures) | 1 | 0
Urinary cystectomy (Surgical and medical procedures) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 13
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma Of The Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal & Squamous Cell Carcinoma's Discovered (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Branchogenic Adenocarcinoma/Right Upper Lobectomy And M (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cytopathology Diagnosis Of Aus/Flus Or Follicular Hurth (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diagnosed With Non Basal Cell Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diagnosis Of Bladder Cancer, Highly Invasive, With Live (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive Squamous Cell Carcinoma (Right Cheek) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Left Descending Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Left Ureteropelvic Junction, Papillary Urothelial Carci (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lesion, Mid-Parietal Scalp, Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liver Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Bladder Polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Spindle Cell Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Transitional Cell Cancer Of The Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Liver Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Micrometastatic Disease Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
New Lung Cancer Diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary Urothelial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peritoneal Carcinomatosis From A Low-Grade Mucinous Tum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pt Newly Diagnosed With Stage 4 Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Recurrent Bladder Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Recurrent Bladder Tumor: Papillary Lesion , Proximal An (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Relapsed Non-Hodgkins Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Reported Diagnosis Lymphoma On Passive Follow Up (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Right Parietal Craniotomy For Benign Neoplasm Of Brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ruptured Mucinous Neoplasm Of The Appendix With Periton (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin Biopsy- Possible Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sqamous Cell Carcinoma In Situ, Bowenoid Type (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Stage Ii Adenocarcinoma Of The Ascending Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Stage Iv T2n0m1 Adenocarcinoma Of Theh Ead And Tail Of (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Treatment For Metastasized Clear Cell Renal Cell Carcin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angina unstable (Cardiac disorders) | 12 | 19
Angina pectoris (Cardiac disorders) | 12 | 6
Bradycardia (Cardiac disorders) | 5 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 7
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 4
Cardiac failure congestive (Cardiac disorders) | 1 | 3
Acute coronary syndrome (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 2
Ventricular fibrillation (Cardiac disorders) | 3 | 0
Arrhythmia (Cardiac disorders) | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery dissection (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pneumopericardium (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 17 | 21
Haematuria (Renal and urinary disorders) | 4 | 4
Nephrolithiasis (Renal and urinary disorders) | 2 | 3
Renal failure (Renal and urinary disorders) | 3 | 2
Renal failure chronic (Renal and urinary disorders) | 3 | 1
Renal mass (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 2
Calculus ureteric (Renal and urinary disorders) | 1 | 1
Bladder mass (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Blood glucose increased (Investigations) | 2 | 5
Catheterisation cardiac (Investigations) | 6 | 1
Arteriogram coronary (Investigations) | 3 | 2
Liver function test abnormal (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 1 | 2
Biopsy bladder (Investigations) | 2 | 0
Stress echocardiogram abnormal (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspiration pleural cavity (Investigations) | 0 | 1
Biopsy breast (Investigations) | 0 | 1
Biopsy liver (Investigations) | 0 | 1
Biopsy lung (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 1 | 0
Bronchoscopy (Investigations) | 0 | 1
Cardiac stress test abnormal (Investigations) | 0 | 1
Cystoscopy (Investigations) | 1 | 0
Haemoglobin increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Hepatitis C virus test positive (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 1
Shift to the right (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 5
Hip fracture (Injury, poisoning and procedural complications) | 4 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Testicular injury (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Traumatic arthropathy (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Obesity (Metabolism and nutrition disorders) | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 7 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (AE & Lab Combined) (Blood and lymphatic system disorders) | 2 | 0 — Data come from laboratory assays and adverse event reports
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (AE & Lab Combined) (Blood and lymphatic system disorders) | 1 | 1 — Data come from laboratory assays and adverse event reports
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukoerythroblastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (AE & Lab Combined) (Blood and lymphatic system disorders) | 1 | 0 — Data come from laboratory assays and adverse event reports
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
White blood cell disorder (Blood and lymphatic system disorders) | 0 | 1
Hypotension (Vascular disorders) | 8 | 3
Hypertension (Vascular disorders) | 2 | 2
Orthostatic hypotension (Vascular disorders) | 4 | 0
Aneurysm (Vascular disorders) | 2 | 1
Aortic stenosis (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 5 | 2
Cholecystitis acute (Hepatobiliary disorders) | 2 | 4
Cholelithiasis (Hepatobiliary disorders) | 3 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Pneumobilia (Hepatobiliary disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 4
Confusional state (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 1
Eye pain (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Any Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 52 | 30 — Reported in case-report forms from visits
Any Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 106 | 95 — Determined on the basis of a MedDRA query, case-report forms from visits and adverse-event reports
Non-basal-cell skin cancer (not known if SAE) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 31 | 10 — Reported in case-report forms from visits
Non-basal-cell skin cancer (not known if SAE) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 33 | 12 — Determined on the basis of a MedDRA query, case-report forms from visits and adverse-event reports
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=2391) | Placebo (N=2395)
Any (Infections and infestations) | 659 | 584 — All diagnoses under the organ system
Any (Gastrointestinal disorders) | 350 | 284 — All diagnoses under the organ system
Any (Blood and lymphatic system disorders) | 340 | 244 — All diagnoses under the organ system
Any (General disorders) | 279 | 254 — All diagnoses under the organ system
Any (Respiratory, thoracic and mediastinal disorders) | 279 | 210 — All diagnoses under the organ system
Any (Musculoskeletal and connective tissue disorders) | 223 | 230 — All diagnoses under the organ system
Any (Investigations) | 220 | 211 — All diagnoses under the organ system
Any (Nervous system disorders) | 213 | 195 — All diagnoses under the organ system
Any (Injury, poisoning and procedural complications) | 150 | 163 — All diagnoses under the organ system
Any (Surgical and medical procedures) | 137 | 147 — All diagnoses under the organ system
Any (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 124 | 101 — All diagnoses under the organ system
Any (Skin and subcutaneous tissue disorders) | 97 | 121 — All diagnoses under the organ system
Leukopenia (Blood and lymphatic system disorders) | 241 | 172 — Data come from laboratory assays and adverse-event reports
Chest pain (General disorders) | 126 | 142

LIMITATIONS AND CAVEATS:
The trial was terminated early because the pre-specified boundary for futility was crossed for both the original and the final primary endpoints and because of the lack of evidence of a reduction in hsCRP level with methotrexate treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT01594333/Prot_SAP_000.pdf